CLINICAL TRIAL: NCT04520425
Title: Osteopathic Manipulative Techniques for the Treatment of Chronic Migraine Headaches
Acronym: SMART-CM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Responsible Party left institution
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00014287
Record Dates: First submitted 2020-08-13; First posted 2020-08-20 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Chronic Migraine, Headache
Keywords: migraine; chronic migraine; osteopathic manipulative therapy
MeSH Terms: conditions — Headache; Migraine Disorders | interventions — Manipulation, Osteopathic; Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: Consenting chronic migraine patients will receive 3-5 standardized osteopathic manipulative treatments over the course of ten weeks, and will be assessed for acceptance and efficacy of the treatment.
Masking Description: As a single arm trial, all participants will know they are receiving a treatment. While the investigator and outcomes assessor will not know which particular patients reported individual responses, they will know that all patients received the same treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants will receive 5 standardized osteopathic manipulative treatments, two weeks apart. (To be considered a study completer, a participant must complete at least 3 of these treatments.) In addition to assessments at intake and during treatments, 1 and 3 months after their last treatment patients will be asked to provide follow-up data. Assessments include the HIT-6, MIDAS, and MSQ surveys, treatment satisfaction assessments, and a headache diary. Participants will also consent to an electronic medical record extraction of medication and healthcare services utilization.
  Interventions: Procedure: Osteopathic manipulative therapy

INTERVENTIONS:
Procedure: Osteopathic manipulative therapy — 1. Mandibular: the clinician applies gentle pressure bilaterally to the subject's mandible, in the direction of the patient's clavicles.
  2. Frontal: the clinician applies gentle pressure bilaterally to the subject's forehead, in a direction halfway between the parietals and ears.
  3. Temporal: the clinician applies gentle pressure bilaterally to the subject's temples, in the direction of the patient's occiput.
  4. Parietal: the clinician applies gentle pressure bilaterally to the subject's parietal bones, in the direction of the patient's occipital atlanto joint.
  5. Occipital: the clinician applies gentle pressure to the subject's occipital bone, in the direction of the patient's neck.
  Other Names: OMT, myofascial release

SUMMARY:
This study evaluates a standardized osteopathic manipulative therapy (OMT) as a treatment for chronic migraine headaches. It will determine the feasibility of enrolling patients in standardized osteopathic manipulative therapy trials, the acceptability of this specific treatment to patients, and evaluate its preliminary effectiveness.

DETAILED DESCRIPTION:
In the United States, 12% of adults suffer from migraines. Migraines are categorized as episodic or chronic (CM). CM is less common than episodic, with a prevalence of 2%, but far more debilitating, with three times the annual per capita cost, putting the total U.S. direct and indirect cost estimate of CM at $15.5 billion dollars per year. Compared to patients with episodic migraine, those with CM have a lower quality of life (QoL) and higher utilization of primary and emergency care. CM has only two prophylactic pharmacologic treatment options with efficacy demonstrated through randomized, placebo-controlled trials. One is Topiramate, whose side effects, including fatigue, dizziness, mood changes and suicidal ideation, can compromise patients' QoL and adherence rate to this treatment, which has been estimated as under 25%. The other is onabotulinumtoxinA, whose side effects, including neck pain, eyelid ptosis and worsening headaches, are reported in over 25% of users. Due to these high frequency, debilitating side effects, ¬there is an urgent need to develop effective CM treatments with low side-effect profiles.

Osteopathic manipulative treatment (OMT) has been reported to improve episodic and CM symptoms without major side effects. Improvements with OMT include decreased Headache Impact Test (HIT-6) scores, fewer headache days per month and decreased medication use. While promising, these studies have significant limitations, such as small sample sizes and high risk of bias. Further, even higher quality OMT studies rely on the treating physician to select from among several OMT treatment techniques, rather than using a standardized treatment procedure. Together, these limitations led the most recent literature assessment to conclude that, "more study is needed before manipulative therapies can be confidently recommended to prevent and treat headaches." To overcome these limitations, OMT studies for the treatment of CM should apply rigorous methods, including standardized treatment procedures.

The investigators have developed a standardized OMT procedure to treat CM. The procedure is repeated every two weeks over a ten week period. Over the past five years it has been successfully used to treat 50 patients with CM in a single family physician's practice. Among the treated patients, 40 reported improved symptoms, and none reported adverse side effects. However, the procedure has not been formally evaluated using rigorous research methods.

The specific objectives of this pilot study are to evaluate the feasibility and acceptability of the standardized OMT procedure for CM, and gather preliminary data on its potential efficacy when implemented in a primary care setting. The central hypothesis is that the standardized myofascial release OMT procedure will improve symptoms of CM as measured by improvement in HIT-6, Migraine Disability Assessment (MIDAS), Migraine-Specific Quality-of-Life Questionnaire (MSQ), and self-reported and electronic health record (EHR) medication usage and healthcare utilization. This hypothesis is supported by the investigators' anecdotal clinical success using this approach. The specific aims of this study are:

Aim 1: Assess the feasibility of systematically identifying and treating patients with the standardized OMT procedure within the Penn State Health medical system. Feasibility will be measured by the investigators' ability to identify and enroll CM patients in this study. The investigators will enroll 20-40 adult patients with CM who do not have common confounders. This data will inform the recruitment strategy of a future randomized clinical trial (RCT).

Aim 2: Assess the acceptability of the standardized OMT procedure. Acceptability will be measured by patient-reported satisfaction and perceived benefit, completion rate and adverse events or side-effects. This data will inform the sample size calculation of a future RCT.

Aim 3: Assess the preliminary effectiveness of the standardized OMT procedure. Efficacy will be measured by improvement in HIT-6, MIDAS, and MSQ scores; patient-reported headache frequency, medication usage, and healthcare utilization surveys; and medication and healthcare utilization documented in the EHR. This data will provide estimates of effect size to better inform the sample size calculation of a future RCT.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study patients must be:

1. An adult ≥ 18 years of age and ≤ 60 years of age
2. Enrolled for care at Penn State Hershey Family and Community Medicine as demonstrated by at least one primary care visit within the past 3 years
3. Diagnosed with chronic migraine (as defined by the International Headache Society: "Headache occurring on 15 or more days/month for more than 3 months, which, on at least 8 days/month, has the features of migraine headache"
4. Legally and physically able to consent in English
5. Willing and able to complete seven in-person visits, each approximately 30 minutes in length, over the course of 21 weeks.

Exclusion Criteria:

Patients will be ineligible to participate in this study if they:

1. Are diagnosed with secondary headache
2. Are pregnant (as reported at the time of enrollment; no pregnancy test is required; patients who become pregnant during the study will be withdrawn from the study. (However, they may continue to receive non-study related OMT treatments through their primary care provider as OMT has been shown to be safe in pregnancy.))
3. Are less than 18 or more than 60 years of age
4. Are diagnosed with fibromyalgia.
5. Have current or prior migraine or other headache treatment with onabotulinumtoxinA (Botox®)
6. Have received any treatment of neck or head with onabotulinumtoxinA (Botox®) within the past year
7. Have current or prior (within 12 months) treatment for any condition with Topiramate
8. Are determined by the physician administering OMT to have a medical condition, history, or medication that is likely to decrease the efficacy or increase the risk of OMT. Not all patients with the following conditions will be excluded, but some patients with any of the following may be determined to be unlikely to benefit from OMT or at increased risk of OMT, and will be excluded.

   1. A history of surgery in the head or neck (except for: uncomplicated dental surgery that is more than 2 years prior and required no significant implantation (i.e., routine wisdom tooth extraction, braces, or root canal))
   2. Unstable mental health disorders
   3. Chronic chronic inflammatory disorders, severe osteoporosis, tumors, evidence of central nervous system pathology include facial palsy, abnormality in vision, speech or balance, paresthesia, or weakness
   4. Have had previous osteopathic treatment for migraine or other headache
   5. Have current or past substance abuse disorder
   6. Have current or pending disability payments, applications for disability or litigation for disability.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Recruitment metrics | 6 months
  Number of eligible patients identified through electronic medical record search, number of contacts needed to schedule an appointment, number of consent meetings to enroll a patient, number of patients who complete the study
Treatment satisfaction, first treatment | 1st treatment, week 12
  5 point Likert-type scale assessing: treatment satisfaction on the day of treatment and likelihood of continuing treatments.
Treatment satisfaction, second treatment | 2nd treatment, week 14
  5 point Likert-type scale assessing: treatment satisfaction on the day of treatment, likelihood of continuing treatments, and (for treatments 2-5) how helpful the treatments have been overall in managing the subjects' chronic migraine
Treatment satisfaction, second treatment | 3rd treatment, week 16
  5 point Likert-type scale assessing: treatment satisfaction on the day of treatment, likelihood of continuing treatments, and (for treatments 2-5) how helpful the treatments have been overall in managing the subjects' chronic migraine
Treatment satisfaction, second treatment | 4th treatment, week 18
  5 point Likert-type scale assessing: treatment satisfaction on the day of treatment, likelihood of continuing treatments, and (for treatments 2-5) how helpful the treatments have been overall in managing the subjects' chronic migraine
Treatment satisfaction, second treatment | 5th treatment, week 20
  5 point Likert-type scale assessing: treatment satisfaction on the day of treatment, likelihood of continuing treatments, and (for treatments 2-5) how helpful the treatments have been overall in managing the subjects' chronic migraine

SECONDARY OUTCOMES:
Headache impact test (HIT-6) | 1st treatment, week 12
  A validated method of measuring headache morbidity
Headache impact test (HIT-6) | 1 month post-intervention, week 24
  A validated method of measuring headache morbidity
Headache impact test (HIT-6) | 3 months post-intervention, week 36
  A validated method of measuring headache morbidity
MIDAS (Migraine Disability Assessment Test) | 1st treatment, week 12
  A validated method of measuring headache morbidity
MIDAS (Migraine Disability Assessment Test) | 3 months post-intervention, week 36
  A validated method of measuring headache morbidity
MSQ (Migraine Specific Quality of Life Questionnaire Version 2.1) | 1st treatment, week 12
  A validated method of measuring headache morbidity
MSQ (Migraine Specific Quality of Life Questionnaire Version 2.1) | 1 month post-intervention, week 24
  A validated method of measuring headache morbidity
MSQ (Migraine Specific Quality of Life Questionnaire Version 2.1) | 3 months post-intervention, week 36
  A validated method of measuring headache morbidity
Headache Diary | 2nd treatment, week 14
  A validated self-assessment method of measuring headache morbidity
Headache Diary | 3rd treatment, week 16
  A validated self-assessment method of measuring headache morbidity
Headache Diary | 4th treatment, week 18
  A validated self-assessment method of measuring headache morbidity
Headache Diary | 5th treatment, week 20
  A validated self-assessment method of measuring headache morbidity
Headache Diary | 1 month post-intervention, week 24
  A validated self-assessment method of measuring headache morbidity
Headache Diary | 3 months post-intervention, week 36
  A validated self-assessment method of measuring headache morbidity
Medication Use | 3 months post-intervention from electronic health record, week 36
  A measurement of total type and amount of medication used to manage migraines, obtained from patient reports on their Headache Diary and from the electronic medical record at the end of the study.
Healthcare Utilization | 3 months post-intervention from electronic health record, week 36
  A measurement of the total type and number of healthcare visits as self reported in the Headache Diary and extracted from the electronic health record at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Lennon, MD, Principal Investigator — Penn State Health Milton S Hershey Medical Center
Locations (1):
- Penn State College of Medicine, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.

REFERENCES:
- [Background] Burch RC, Buse DC, Lipton RB. Migraine: Epidemiology, Burden, and Comorbidity. Neurol Clin. 2019 Nov;37(4):631-649. doi: 10.1016/j.ncl.2019.06.001. Epub 2019 Aug 27. PMID 31563224
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Messali A, Sanderson JC, Blumenfeld AM, Goadsby PJ, Buse DC, Varon SF, Stokes M, Lipton RB. Direct and Indirect Costs of Chronic and Episodic Migraine in the United States: A Web-Based Survey. Headache. 2016 Feb;56(2):306-22. doi: 10.1111/head.12755. Epub 2016 Feb 1. PMID 26833083
- [Background] Bonafede M, Sapra S, Shah N, Tepper S, Cappell K, Desai P. Direct and Indirect Healthcare Resource Utilization and Costs Among Migraine Patients in the United States. Headache. 2018 May;58(5):700-714. doi: 10.1111/head.13275. Epub 2018 Feb 15. PMID 29446063
- [Background] Diener HC, Solbach K, Holle D, Gaul C. Integrated care for chronic migraine patients: epidemiology, burden, diagnosis and treatment options. Clin Med (Lond). 2015 Aug;15(4):344-50. doi: 10.7861/clinmedicine.15-4-344. PMID 26407383
- [Background] Silberstein SD. Topiramate in Migraine Prevention: A 2016 Perspective. Headache. 2017 Jan;57(1):165-178. doi: 10.1111/head.12997. Epub 2016 Nov 30. PMID 27902848
- [Background] Chiang CC, Starling AJ. OnabotulinumtoxinA in the treatment of patients with chronic migraine: clinical evidence and experience. Ther Adv Neurol Disord. 2017 Dec;10(12):397-406. doi: 10.1177/1756285617731521. Epub 2017 Sep 20. PMID 29204191
- [Background] Cerritelli F, Ginevri L, Messi G, Caprari E, Di Vincenzo M, Renzetti C, Cozzolino V, Barlafante G, Foschi N, Provinciali L. Clinical effectiveness of osteopathic treatment in chronic migraine: 3-Armed randomized controlled trial. Complement Ther Med. 2015 Apr;23(2):149-56. doi: 10.1016/j.ctim.2015.01.011. Epub 2015 Jan 21. PMID 25847552
- [Background] Smith MS, Olivas J, Smith K. Manipulative Therapies: What Works. Am Fam Physician. 2019 Feb 15;99(4):248-252. PMID 30763049
- [Background] Chaibi A, Tuchin PJ, Russell MB. Manual therapies for migraine: a systematic review. J Headache Pain. 2011 Apr;12(2):127-33. doi: 10.1007/s10194-011-0296-6. Epub 2011 Feb 5. PMID 21298314
- [Background] Chaibi A, Benth JS, Tuchin PJ, Russell MB. Chiropractic spinal manipulative therapy for migraine: a three-armed, single-blinded, placebo, randomized controlled trial. Eur J Neurol. 2017 Jan;24(1):143-153. doi: 10.1111/ene.13166. Epub 2016 Oct 2. PMID 27696633
- [Background] Voigt K, Liebnitzky J, Burmeister U, Sihvonen-Riemenschneider H, Beck M, Voigt R, Bergmann A. Efficacy of osteopathic manipulative treatment of female patients with migraine: results of a randomized controlled trial. J Altern Complement Med. 2011 Mar;17(3):225-30. doi: 10.1089/acm.2009.0673. Epub 2011 Mar 8. PMID 21385086
- [Background] Park PW, Dryer RD, Hegeman-Dingle R, Mardekian J, Zlateva G, Wolff GG, Lamerato LE. Cost Burden of Chronic Pain Patients in a Large Integrated Delivery System in the United States. Pain Pract. 2016 Nov;16(8):1001-1011. doi: 10.1111/papr.12357. Epub 2015 Oct 7. PMID 26443292
- [Background] GBD 2016 Headache Collaborators. Global, regional, and national burden of migraine and tension-type headache, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2018 Nov;17(11):954-976. doi: 10.1016/S1474-4422(18)30322-3. PMID 30353868
- [Background] Stevinson C, Ernst E. Risks associated with spinal manipulation. Am J Med. 2002 May;112(7):566-71. doi: 10.1016/s0002-9343(02)01068-9. PMID 12015249
- [Background] Hayes NM, Bezilla TA. Incidence of iatrogenesis associated with osteopathic manipulative treatment of pediatric patients. J Am Osteopath Assoc. 2006 Oct;106(10):605-8. PMID 17122030
- [Background] Odell J, Clark C, Hunnisett A, Ahmed OH, Branney J. Manual therapy for chronic migraine: a pragmatic randomised controlled trial study protocol. Chiropr Man Therap. 2019 Mar 27;27:11. doi: 10.1186/s12998-019-0232-4. eCollection 2019. PMID 30962877
- [Background] Hensel KL, Carnes MS, Stoll ST. Pregnancy Research on Osteopathic Manipulation Optimizing Treatment Effects: The PROMOTE Study Protocol. J Am Osteopath Assoc. 2016 Nov 1;116(11):716-724. doi: 10.7556/jaoa.2016.142. PMID 27802557
- [Background] Coeytaux RR, Kaufman JS, Chao R, Mann JD, Devellis RF. Four methods of estimating the minimal important difference score were compared to establish a clinically significant change in Headache Impact Test. J Clin Epidemiol. 2006 Apr;59(4):374-80. doi: 10.1016/j.jclinepi.2005.05.010. PMID 16549259
- [Background] Hammond NG, Stinchcombe A. Health Behaviors and Social Determinants of Migraine in a Canadian Population-Based Sample of Adults Aged 45-85 Years: Findings From the CLSA. Headache. 2019 Oct;59(9):1547-1564. doi: 10.1111/head.13610. Epub 2019 Aug 2. PMID 31373683
- [Background] Yang M, Rendas-Baum R, Varon SF, Kosinski M. Validation of the Headache Impact Test (HIT-6) across episodic and chronic migraine. Cephalalgia. 2011 Feb;31(3):357-67. doi: 10.1177/0333102410379890. Epub 2010 Sep 6. PMID 20819842
- [Background] Rendas-Baum R, Yang M, Varon SF, Bloudek LM, DeGryse RE, Kosinski M. Validation of the Headache Impact Test (HIT-6) in patients with chronic migraine. Health Qual Life Outcomes. 2014 Aug 1;12:117. doi: 10.1186/s12955-014-0117-0. PMID 25080874
- [Background] Stewart WF, Lipton RB, Dowson AJ, Sawyer J. Development and testing of the Migraine Disability Assessment (MIDAS) Questionnaire to assess headache-related disability. Neurology. 2001;56(6 Suppl 1):S20-8. doi: 10.1212/wnl.56.suppl_1.s20. PMID 11294956
- [Background] Rendas-Baum R, Bloudek LM, Maglinte GA, Varon SF. The psychometric properties of the Migraine-Specific Quality of Life Questionnaire version 2.1 (MSQ) in chronic migraine patients. Qual Life Res. 2013 Jun;22(5):1123-33. doi: 10.1007/s11136-012-0230-7. Epub 2012 Jul 15. PMID 22797868
- [Background] Cole JC, Lin P, Rupnow MF. Minimal important differences in the Migraine-Specific Quality of Life Questionnaire (MSQ) version. Cephalalgia. 2009 Nov;29(11):1180-7. doi: 10.1111/j.1468-2982.2009.01852.x. PMID 19830883
- [Background] Jensen R, Tassorelli C, Rossi P, Allena M, Osipova V, Steiner T, Sandrini G, Olesen J, Nappi G; Basic Diagnostic Headache Diary Study Group. A basic diagnostic headache diary (BDHD) is well accepted and useful in the diagnosis of headache. a multicentre European and Latin American study. Cephalalgia. 2011 Nov;31(15):1549-60. doi: 10.1177/0333102411424212. Epub 2011 Oct 21. PMID 22019575
- [Background] Bigal ME, Serrano D, Reed M, Lipton RB. Chronic migraine in the population: burden, diagnosis, and satisfaction with treatment. Neurology. 2008 Aug 19;71(8):559-66. doi: 10.1212/01.wnl.0000323925.29520.e7. PMID 18711108